CLINICAL TRIAL: NCT02194322
Title: A Double-blind (at Each Dose Level), Randomised, Placebo-controlled Single Increasing Dose Safety, Tolerability and Pharmacokinetics Study in Healthy Male and Female Volunteers After Intranasal Administration of BIBN 4096 BS (Dosage: 6.25 mg - 200mg )
Brief Title: Safety, Tolerability and Pharmacokinetics After Administration of Increasing Dose of BIBN 4096 BS in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1149.35
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BIBN 4096 BS - in single rising doses (Experimental)
  Interventions: Drug: BIBN 4096 BS - in single rising doses
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIBN 4096 BS - in single rising doses
  Arms: BIBN 4096 BS - in single rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of the present study is to obtain information about the safety, tolerability and pharmacokinetics of BIBN 4096 BS after single intranasal administration of increasing doses in healthy male and female volunteers

ELIGIBILITY:
Inclusion Criteria:

* Participants should be healthy males and females
* Age range from 21 to 50 years
* Body Mass Index (BMI) is to be within 18.5 to 29.9 kg/m² (BMI calculation: weight in kilograms divided by the square of height in meters)
* In accordance with Good Clinical Practice (GCP) and local legislation each volunteers are supposed to give their written informed consent prior to admission to the study
* As part of the screening (within 14 days before drug administration), each subject was to receive a complete medical examination (including blood pressure, pulse rate, medical history, documentation of demographics, inclusion/exclusion criteria and concomitant therapy) as well as a 12-lead Electrocardiogram (ECG) and a rhinomanometry (in order to familiarize the subject with this method; screening rhinomanometric values were not to be reported). Moreover laboratory parameters (including drug screening, HBs- antigen (HBs-Ag), anti Hepatitis B core (HBc) - antibodies, anti Hepatitis C Virus (HCV) - antibodies and Human immunodeficiency virus (HIV) test as well as pregnancy test for female subjects are to be determined.

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or with psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of a drug with a long half-life (> 24 hours) within at least 1 month or less than ten half-lives of the respective drug before enrolment in the study (except substitution therapy regarding thyroid gland/or ovaries)
* Use of any drugs which might influence the results of the trial within 1 week prior to administration or during the trial
* Participation in another study with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse (> 60g/day)
* Drug abuse
* Blood donation (>= 100 ml) within four weeks prior to administration or during the trial
* Excessive physical activities within the last week before the study
* Any laboratory value outside the reference range of clinical relevance

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. oral contraceptives, sterilization, intrauterine pessary (IUP)
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2001-11; Primary Completion 2002-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 24 days
Number of patients with abnormal changes in laboratory parameters | up to 24 days
Number of patients with clinically significant changes in vital signs (blood pressure, pulse rate) | up to 24 days
Number of patients with clinically significant changes in 12-lead Electrocardiogram (ECG) | up to 24 days
Assessment of tolerability on a 4-point scale | 8 days after drug administration
Macroscopic changes in nasal mucosa assessed by rhinoscopy | up to 3 hours after drug administration
Changes in nasal flow assessed by rhinomanometry | up to 3 hours after drug administration

SECONDARY OUTCOMES:
Cmax (Maximum measured concentration of the analyte in plasma) | up to 48 hours after drug administration
tmax (Time from dosing to the maximum concentration of the analyte in plasma) | up to 48 hours after drug administration
AUC0-tz (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | up to 48 hours after drug administration
AUC0-∞ (Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 48 hours after drug administration
t½ (Terminal half-life of the analyte in plasma) | up to 48 hours after drug administration
λz (Terminal rate constant in plasma) | up to 48 hours after drug administration
CL/F (Apparent clearance of the analyte in plasma following extravascular administration) | up to 48 hours after drug administration
MRTtot (Total mean residence time of the analyte) | up to 48 hours after drug administration
Vz/F (Apparent volume of distribution of the analyte during the terminal phase) | up to 48 hours after drug administration
CLR (Renal clearance of the analyte in plasma) | up to 48 hours after drug administration
Ae (Amount of parent drug excreted into urine) | up to 24 hours after drug administration